CLINICAL TRIAL: NCT00002442
Title: A Phase II, Open-Label, Randomized Study of the Efficacy and Safety of Epivir 150 Mg BID Versus Epivir 300 Mg Once-Daily When Administered for 24 Weeks in Combination With FDA-Approved Dosage Regimens of Zerit and Either Crixivan or Viracept in Subjects With HIV-1 Infection
Brief Title: A Study to Compare the Safety and Effectiveness of Two Dosing Schedules of Lamivudine in Combination With Two Other Anti-HIV Drugs
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Glaxo Wellcome (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Masking: None | Purpose: Treatment
Other Study IDs: 225C; COLA 4005
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2000-08

CONDITIONS: HIV Infections
Keywords: Drug Therapy, Combination; Zidovudine; Drug Administration Schedule; Stavudine; HIV Protease Inhibitors; Lamivudine; Indinavir; Dosage Forms; Nelfinavir; Reverse Transcriptase Inhibitors; Anti-HIV Agents
MeSH Terms: conditions — HIV Infections | interventions — Indinavir; Nelfinavir; Lamivudine; Stavudine

INTERVENTIONS:
Drug: Indinavir sulfate
Drug: Nelfinavir mesylate
Drug: Lamivudine
Drug: Stavudine

SUMMARY:
The purpose of this study is to compare the safety and effectiveness of 2 dosing schedules (once daily vs twice daily) of lamivudine (3TC) given with stavudine (d4T) and either indinavir (IDV) or nelfinavir (NFV) for 24 weeks.

DETAILED DESCRIPTION:
Patients are randomized to 1 of 2 groups. Group 1 receives 3TC qd plus d4T plus either IDV or NFV. Group 2 receives 3TC bid plus d4T plus either IDV or NFV. Patients are evaluated for drug tolerance, medication adherence, and genotypic and phenotypic resistance.

ELIGIBILITY:
Inclusion Criteria

Patients may be eligible for this study if they:

* Are HIV-positive.
* Are at least 18 years old.
* Have had an HIV level below 400 copies/ml for at least 3 months prior to study entry.
* Have a CD4 cell count of at least 50 cells/mm3.
* Are currently taking an anti-HIV drug regimen that includes 3TC plus d4T plus either IDV or NFV for at least 6 months prior to study entry. (Note: This must be their first anti-HIV drug regimen.)
* Agree to abstain from sex or use effective methods of birth control during the study.

Exclusion Criteria

Patients will not be eligible for this study if they:

* Have a history of an AIDS-defining illness or certain other medical conditions.
* Are allergic to any of the study drugs.
* Are unable to take medication by mouth for any reason.
* Have received certain medications.
* Will need to receive radiation therapy or chemotherapy (for any cancer other than Kaposi's sarcoma) during the study.
* Are pregnant or breast-feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1999-06

CONTACTS AND LOCATIONS:
Locations (12):
- United States (12):
  - AIDS Healthcare Foundation, Los Angeles, California
  - Palo Alto Veterans Affairs Health Care System, Palo Alto, California
  - Dupont Circle Physicians Group, Washington D.C., District of Columbia
  - IDC Research Initiative, Altamonte Springs, Florida
  - North Broward Hosp District, Fort Lauderdale, Florida
  - Steinhart Medical Associates, Miami, Florida
  - Northwestern Univ Med School, Chicago, Illinois
  - Saint Vincents Hosp, New York, New York
  - St Lukes - Roosevelt Hosp Ctr, New York, New York
  - MCP Hahnemann Univ Hosp, Philadelphia, Pennsylvania
  - Southwest Infectious Disease Association / PA, Dallas, Texas
  - Univ TX Galveston Med Branch, Galveston, Texas